CLINICAL TRIAL: NCT03625310
Title: Effectiveness of Different Fluoride Varnishes on Salivary Bacteria Levels in Children With Early Childhood Caries
Brief Title: Effectiveness Fluoride Varnishes in Children With Early Childhood Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merve Erkmen Almaz (Other)
Responsible Party: Sponsor-Investigator, Merve Erkmen Almaz, assist prof, Kırıkkale University
Organization: Kırıkkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Kirikkale University
Record Dates: First submitted 2018-07-27; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Early Childhood Caries
MeSH Terms: interventions — Sodium Fluoride; tenocyclidine; casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sodium Fluoride (Active Comparator): Varnish containing 5% Sodium Fluoride, was applied to all remaining teeth of each child after dental treatment under general anaesthesia.
  Interventions: Drug: Sodium Fluoride
- Sodium Fluoride with TCP (Experimental): Varnish containing 5% Sodium Fluoride with tricalcium phosphate (TCP) ,varnish was applied to all remaining teeth of each child after dental treatment under general anaesthesia.
  Interventions: Drug: Sodium Fluoride with TCP
- Sodium Fluoride with CXP (Experimental): Varnish containing 5% Sodium Fluoride with Xylitol-coated Calcium and Phosphate (CXP) ,varnish was applied to all remaining teeth of each child after dental treatment under general anaesthesia.
  Interventions: Drug: Sodium Fluoride with CXP
- Sodium Fluoride with CPP-ACP (Experimental): Varnish containing 5% Sodium Fluoride with casein phosphopeptide amorphous calcium phosphate (CPP-ACP), varnish was applied to all remaining teeth of each child after dental treatment under general anaesthesia.
  Interventions: Drug: Sodium Fluoride with CPP-ACP

INTERVENTIONS:
Drug: Sodium Fluoride
  Other Names: Colgate Duraphat varnish
  Arms: Sodium Fluoride
Drug: Sodium Fluoride with TCP
  Other Names: Clinpro ™ White Varnish 3M ESPE
  Arms: Sodium Fluoride with TCP
Drug: Sodium Fluoride with CXP
  Other Names: Embrace ™ Varnish Pulpdent
  Arms: Sodium Fluoride with CXP
Drug: Sodium Fluoride with CPP-ACP
  Other Names: MI Varnish GC
  Arms: Sodium Fluoride with CPP-ACP

SUMMARY:
The study was carried out in 88 children with severe early childhood caries (dmfs≥age +1) who were referred to the investigators' clinic. Patients who completed dental treatment under general anesthesia in a single session, were included to the study.

Patients were divided randomly into 4 groups and after dental treatment one of the fluoride varnish listed below was applied to each child. The groups were as follows;

1. Duraphat varnish containing 5% Sodium Fluoride (Colgate) (n = 22),
2. Clinpro ™ White Varnish containing 5% of Sodium Fluoride tricalcium phosphate (3M ESPE) (n = 22),
3. Embrace ™ Varnish containing 5% Sodium Fluoride with CXP ™ (Pulpdent) (n = 22),
4. MI Varnish containing 5% Sodium Fluoride casein phosphopeptide amorphous calcium phosphate varnish (GC) (n = 22).

Saliva Mutans streptococci (MS) and Lactobacilli (LB) levels, were evaluated by taking saliva samples before general anaesthesia; one month after treatment and three months after treatment.

DETAILED DESCRIPTION:
Duraphat (Colgate), which we used as a positive control group in our study, contains only 5% sodium fluoride. It has been reported in studies that Duraphat is effective in remineralization.

Clinpro ™ White Varnish, another topical varnish in this study,was reported to be effective for caries prevention in pre-school children.

One of the varnishes we evaluate in the study, Embrace™ Varnish, contains 5% sodium fluoride with xylitol-coated calcium and phosphate. According to the manufacturer, the xylitol coating prevents the calcium and phosphate salts from reacting until they come in contact with saliva. Saliva dissolves the xylitol and releases the calcium and phosphate ions, which react with the fluoride ions in saliva to form protective fluorapatite on the teeth19 MI Varnish, in the fourth group containing 5% sodium fluoride with casein phosphopeptide amorphous calcium phosphate (CPP-ACP) had a high release of calcium and fluoride ions.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of healthy children with severe early childhood caries,
* younger than 6 years in the primary dentition

Exclusion Criteria:

* history of any chronic disease,
* use of any drugs that reduce salivary flow or antibiotics in the last 4 weeks,
* use of systemic fluoride tablets

Ages: 36 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Effect of fluoride varnishes on saliva Mutans streptococci (MS) and Lactobacilli (LB) levels were evaluated as colony forming units (CFU). | 3 months
  Saliva Mutans streptococci (MS) and Lactobacilli (LB) levels, were evaluated by taking saliva samples using CRT Bacteria (Caries Risk Test, Ivoclar Vivadent)

REFERENCES:
- [Derived] Erkmen Almaz M, Akbay Oba A. Antibacterial activity of fluoride varnishes containing different agents in children with severe early childhood caries: a randomised controlled trial. Clin Oral Investig. 2020 Jun;24(6):2129-2136. doi: 10.1007/s00784-020-03300-w. Epub 2020 Apr 30. PMID 32356211